CLINICAL TRIAL: NCT03241537
Title: Open Label, Randomized Phase III Trial of Hormone Therapy Alone Versus COmbined HOrmone With Radiation Therapy in Clinical Pelvic Lymph Node Metastatic Prostate Cancer (COHORT Trial)
Brief Title: COHORT Trial in Clinical Pelivc Lymph Node Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC2015-11-139-002
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hormonal therapy alone (No Intervention): total androgen ablation or antiandrogen therapy alone for 2-3 years
- Hormonal therapy with radiotherapy (Active Comparator): total androgen ablation or antiandrogen therapy for 2-3 years combined with radiotherapy on whole pelvis
  Interventions: Radiation: Intensity modulated radiotherapy

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy
  Arms: Hormonal therapy with radiotherapy

SUMMARY:
In local advanced prostate cancer patients with clinically positive metastatic regional lymph node, the optimal treatment is still unanswered. For these patients, radiotherapy combined with hormonal therapy or hormonal therapy alone are recommended. Recently, the reports from NCCB and SEER data showed that radiotherapy combined with hormonal therapy have better survivals than hormonal therapy alone.

This randomized phase III trial compare hormonal therapy alone with combined hormone with radiotherapy in clinically pelvic lymph node metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed prostate cancer within 6 months for study enrollment
* Clincally enlarged pelvic lymph node ((short axis 0.5 cm ≤) in imaging studies (CT, MRI, PET-CT) at diagnosis and partial response or complete remission of enlarged lymph nodes according to RECIST v1.1 after hormonal therapy for 2-3 months 3. age 20 ≤ 4. ECOG performance status 0-1 5. Optimal hematologic profiles within 6 months for study enrollment
* Absolute neutrophil count (ANC) ≥ 1500 cells/mm3
* Platelets ≥ 50,000 cells/mm3
* Hemoglobin ≥ 8.0 g/dl 6. Optimal kidney function within 6 months for study enrollment
* Creatinine < 2.0 ng/dL 7. Optimal liver functions within 6 months for study enrollment
* total bilirubin < 1.5 X maximum normal value
* alanine aminotransferase or aspartate aminotransferase < 2.5 X maximum normal value

Exclusion Criteria:

1. combined with distant metastasis (retroperitoneal lymph node, bone,...)
2. previous history of antiandrogen therapy within 6 months of study enrollment
3. previous history of definitive prostate cancer treatment such as prostatectomy
4. previous history of pelvic radiotherapy
5. previous history of other cancer treatment except for skin cancer and theroid cancer

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Comparison of recurrence-free survival between two treatment groups | 5-year
  expected 5-year recurrence-free survival were 40% in hormonal therapy alone group and more than 80% in hormonal therapy combined with radiotherapy

SECONDARY OUTCOMES:
Comparison of toxicities between two treatment groups | 5-year
  Compare adverse events accroding to CTCAE V4.0 between hormonal therapy alone group and hormonal therapy combined with radiotherapy group
Comparison of quality of lifl between two treatment groups | 5-year
  Compare quality of life accroding to Expanded prostate cancer index composite_Korean between hormonal therapy alone group and hormonal therapy combined with radiotherapy group
Comparison of overall survival between two treatment groups | 5-year
  Compare overall survival between hormonal therapy alone group and hormonal therapy combined with radiotherapy group
Comparison of clinical failure free survival between two treatment groups | 5-year
  Compare clinical failure free survival between hormonal therapy alone group and hormonal therapy combined with radiotherapy group
Comparison of cause-specific survival between two treatment groups | 5-year
  Compare cause-specific survival between hormonal therapy alone group and hormonal therapy combined with radiotherapy group

CONTACTS AND LOCATIONS:
Overall Officials: Won Park, M.D.,Ph.D, Principal Investigator — Korean Radiation Oncology Group
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No